CLINICAL TRIAL: NCT02481505
Title: Spinal Anaesthesia With Chloroprocaine HCl 1% for Elective Lower Limb Procedures of Short Duration: a Prospective, Randomised, Observer-blind Study in Adult Patients
Brief Title: Spinal Anaesthesia With Chloroprocaine HCl 1% for Elective Lower Limb Procedures of Short Duration.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Collaborators: Cross S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHL.1/02-2014; 2014-003778-17 (EudraCT Number)
Record Dates: First submitted 2015-06-02; First posted 2015-06-25 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Short Duration Lower Limb Surgery Via Spinal Anaesthesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 mL Chloroprocaine HCl 1% (Experimental): Patients in D1 group will receive a single dose of 3 mL Chloroprocaine HCl 1% (corresponding to 30 mg chloroprocaine HCl)
  Interventions: Drug: Chloroprocaine HCl 1%
- 4 mL Chloroprocaine HCl 1% (Experimental): Patients in D2 group will receive a single dose of 4 mL Chloroprocaine HCl 1% (corresponding to 40 mg chloroprocaine HCl)
  Interventions: Drug: Chloroprocaine HCl 1%
- 5 mL Chloroprocaine HCl 1% (Experimental): Patients in D3 group will receive a single dose of 5 mL Chloroprocaine HCl 1% (corresponding to 50 mg chloroprocaine HCl)
  Interventions: Drug: Chloroprocaine HCl 1%

INTERVENTIONS:
Drug: Chloroprocaine HCl 1% — Intrathecal Route
  Other Names: Ampres 1%

SUMMARY:
This study evaluate the effect of 3 doses of Chloroprocaine HCl 1% (30, 40 and 50 mg) for spinal anaesthesia in adult patients undergoing short duration elective surgery of the lower limb. Patients undergoing elective short-duration lower limb surgery will be randomised into 3 treatment groups (15 patients per group) to receive one of the 3 single doses of Chloroprocaine HCl 1%, i.e. either D1, D2 or D3, via intrathecal injection.

DETAILED DESCRIPTION:
To evaluate the efficacy of the three Chloroprocaine HCl 1% doses (i.e. D1, D2 and D3) in terms of time to complete regression of spinal block (i.e. end of anaesthesia)

ELIGIBILITY:
Inclusion Criteria:

1. Sex, age and surgery: male/female patients, 18-65 years old, scheduled for short duration (less than 40 min) lower limb surgery requiring ≥ T12 metameric level of sensory block
2. Body Mass Index (BMI): 18 - 32 kg/m2 inclusive
3. ASA physical status: I-II
4. Informed consent: signed written informed consent before inclusion in the study 5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study. Contraindications to spinal anaesthesia. History of neuromuscular diseases to the lower extremities
2. ASA physical status: III-V
3. Further anaesthesia: patients expected to require further anaesthesia
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations ingredients; ascertained or presumptive hypersensitivity to the ester type and major anaesthetics
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; ascertained psychiatric and neurological diseases, sepsis, blood coagulation disorders, severe cardiopulmonary disease, thyroid disease, diabetes or other neuropathies.
6. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study, calculated from the first day of the month following the last visit of the previous study
7. Drug, alcohol: history of drug or alcohol abuse
8. Blood donation: blood donations in the 3 months before this study
9. Pregnancy and lactation: missing or positive pregnancy test at screening, pregnant or lactating women
10. Chronic pain syndromes: patients with chronic pain syndromes (taking opioids, antidepressants, anticonvulsant agents or chronic analgesic therapy) 11. Medications: medication known to interfere with the extent of spinal blocks for 2 weeks before the start of the study. Hormonal contraceptives for females are allowed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano MD Bonarelli, Principal Investigator — Istituto Ortopedico Rizzoli, SC Anestesia e Terapia Intensiva post-operatoria e del dolore IOR-IRCCS
Locations (1):
- Stefano Bonarelli, Bologna, Italy

REFERENCES:
- [Derived] Ghisi D, Boschetto G, Spinelli AM, Giannone S, Frugiuele J, Ciccarello M, Bonarelli S. Spinal anaesthesia with Chloroprocaine HCl 1% for elective lower limb procedures of short duration: a prospective, randomised, observer-blind study in adult patients. BMC Anesthesiol. 2021 Feb 20;21(1):58. doi: 10.1186/s12871-021-01279-9. PMID 33610175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1% | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0.0 | 0.0 | 0.0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (11.7) | 39.4 (12.5) | 41.5 (13.9) | 40.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 9 | 9 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Italy | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Time to Regression of Spinal Block
Description: When Bromage score returns to 0 and sensitive perception returns to S1 To evaluate the efficacy of the three Chloroprocaine HCI 1% doses (i.e. 30 mg, 40 mg e 50 mg) in terms of time to complete regression of spinal block (i.e. end of anaesthesia) Bromage Score is comprised between 1 and 4 (1 equals Free movement of legs and feet while 4 stands for Unable to move legs or feet)
Time Frame: Up to 5 hours after regression of two dermatomers
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
minutes | 40.8 (12.1) | 39.4 (12.5) | 41.5 (13.9)

2. Secondary Outcome: Time to Onset of Sensory Block (Corresponding to Readiness for Surgery)
Description: Time period from spinal injection (time 0 h) to achievement of sensory block The evolution of both sensory and motor blocks, including sensory block metameric level, will be evaluated every 2 min until readiness for surgery, every 5 min until the maximum level is reached (two consecutive observations with the same level of sensory block) and then every 5 min until regression of two dermatomers with respect to the maximum level of sensory block.
Time Frame: Up to 40 min after spinal injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
minutes | 5.4 (3) | 6.6 (3.4) | 4.8 (2)

3. Secondary Outcome: Time to Onset of Motor Block
Description: Time period from spinal injection (time 0 h) to achievement of motor block
Time Frame: Up to 40 min after spinal injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
minutes | 6.3 (3.2) | 6 (3.3) | 4.4 (2.3)

4. Secondary Outcome: Time to Readiness for Surgery
Description: Time period from completion of spinal injection (time 0 h) to achievement of sensory and motor block adequate for surgery, i.e. loss of Pinprick sensation and Bromage's score ≥ 2 at the required metameric level ≥ T12
Time Frame: Up to 40 min after spinal injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
minutes | 8 (4.1) | 7.9 (4.7) | 5.3 (2)

5. Secondary Outcome: Time to Regression of Spinal Block
Time Frame: Up to 1 h and 40 min after readiness for surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 1.761 (0.348) | 2.127 (0.457) | 2.229 (0.379)

6. Secondary Outcome: Time to Resolution of Sensory Block to S1(Min)
Description: Time period from spinal injection (time 0 h) to the time when sensitive perception has returned to S1
Time Frame: Up to 5 h after regression of two dermatomers
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 1.761 (0.348) | 2.127 (0.457) | 2.195 (0.386)

7. Secondary Outcome: Time to Resolution of Motor Block
Description: Time period from spinal injection (time 0 h) to the time when the Bromage score has returned to 0 (Bromage Scale comprises from 1 to 4, where 1 equals Free movement of legs and feet while 4 stands for Unable to move legs or feet)
Time Frame: Up to 5 h after regression of two dermatomers
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 2.662 (0.789) | 3.361 (1.120) | 3.213 (0.856)

8. Secondary Outcome: Time to Unassisted Ambulation
Description: Time period from spinal injection (time 0 h) to the time when the patient can walk unassisted
Time Frame: Up to 5 h after regression of two dermatomers
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 2.662 (0.789) | 3.361 (1.120) | 3.213 (0.856)

9. Secondary Outcome: Sensory Block Metameric Level
Description: Metameric level of sensory block assessed from spinal injection (time 0 h) until regression of sensory block to S1
Time Frame: Up to 5 h after regression of two dermatomers
Measure: Number; unit: participants
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
participants
  T2 | 0 | 2 | 2
  T3 | 1 | 0 | 1
  T4 | 3 | 2 | 1
  T6 | 0 | 1 | 4
  T7 | 1 | 0 | 1
  T8 | 3 | 3 | 2
  T10 | 3 | 1 | 3
  T12 | 3 | 5 | 1
  L1 | 1 | 1 | 0

10. Secondary Outcome: Maximum Level of Sensory Block
Description: Maximum metameric level of sensory block (decreased or absent sensation) achieved
Time Frame: Up to 1 h and 40 min after readiness for surgery
Measure: Number; unit: participants
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
participants
  T2 | 0 | 2 | 2
  T3 | 1 | 0 | 1
  T4 | 3 | 2 | 1
  T6 | 0 | 1 | 4
  T7 | 1 | 0 | 1
  T8 | 3 | 3 | 2
  T10 | 3 | 1 | 3
  T12 | 3 | 5 | 1
  L1 | 1 | 1 | 0

11. Secondary Outcome: Time to Maximum Level of Sensory Block
Description: Time period from spinal injection (Tsp; time 0 h) to the time when the maximum metameric level of sensory block is achieved (consider the time of the first of the two consecutive observations with the same level of sensory block)
Time Frame: Up to 1 h and 40 min after readiness for surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
minutes | 0.224 (0.14) | 0.235 (0.077) | 0.234 (0.098)

12. Secondary Outcome: Time to Regression of Two Dermatomers With Respect to the Maximum Level of Sensory Block
Description: Time period from spinal injection (time 0 h) to the time when the sensory block decrease of two dermatomers with respect to the maximum level of sensory block
Time Frame: Up to 5 h after regression of two dermatomers
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 0.687 (0.361) | 0.851 (0.468) | 0.695 (0.290)

13. Secondary Outcome: Time to Eligibility for Home Discharge
Description: Time period from spinal injection (time 0 h) to the time when the criteria from discharge are met, even if according to the hospital procedures the patient is discharged at a later time
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 3.021 (1.012) | 3.545 (1.281) | 3.530 (0.887)

14. Secondary Outcome: Time to First Spontaneous Urine Voiding
Description: Time period from spinal injection ( time 0 h) to the first time when the patient can pass urine unassisted
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 2.530 (0.761) | 3.361 (1.120) | 3.067 (0.755)

15. Secondary Outcome: Time to First Post-operative Analgesia
Description: Time from spinal injection (time 0 h) to first post-operative analgesia
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 8.186 (10.815) | 2.928 (1.228) | 2.988 (1.167)

16. Secondary Outcome: Time to Administration of Rescue Anaesthesia or Rescue Analgesia
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
hours | 0.717 (0.397) | 0.315 (0.049) | 0 (0)

17. Secondary Outcome: Concentration of 2-chloro-4-aminobenzoic Acid (CABA) in Plasma
Time Frame: at pre-dose, 5, 10, 30 and 60 min after spinal puncture
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
minutes
  5 minutes post-dose | 16.127 (20.108) | 20.411 (23.037) | 24.887 (20.340)
  10 minutes post-dose | 41.440 (31.778) | 38.851 (25.492) | 75.833 (67.635)
  30 minutes post-dose | 57.459 (43.773) | 67.180 (36.899) | 97.647 (61.704)
  60 minutes post-dose | 47.020 (41.381) | 53.093 (31.803) | 78.380 (48.403)

18. Secondary Outcome: Excretion of 2-chloro-4-aminobenzoic Acid (CABA) in Urine
Description: Time period from spinal injection ( time 0 h) to the first time when the patient can pass urine unassisted
Time Frame: at the time of first urine voiding post surgery
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
ng/mL | 1217.7 (627.8) | 1827.9 (904.1) | 2103.5 (1537.5)

19. Secondary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: All AEs occurring or worsening after the dose of IMP
Time Frame: Up to Day 6 +/- 1 after spinal puncture
Measure: Number; unit: participants
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
participants
  Procedural pain | 14 | 13 | 13
  Injection site pain | 2 | 3 | 3
  nausea | 0 | 1 | 1
  diarrhea | 0 | 1 | 0
  vomiting | 0 | 1 | 0
  bradycardia | 0 | 1 | 0

20. Secondary Outcome: Transient Neurological Symptoms (TNS)
Time Frame: Up to Day 6 +/- 1 after spinal puncture
Measure: Number; unit: participants
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
participants
  day 2 | 0 | 0 | 0
  day 7 | 0 | 0 | 0

21. Secondary Outcome: Pain Assessment at the Site of Injection and at the Site of Surgery
Description: Number of patients with pain at the site of injection and at the site of surgery
Time Frame: Up to Day 6 +/- 1 after spinal puncture
Measure: Number; unit: participants
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
participants
  Immediately after regression of spinal block | 0 | 0 | 0
  discharge | 0 | 0 | 0
  day 2 | 14 | 15 | 15
  day 7 | 15 | 15 | 15

22. Secondary Outcome: Heart Rate
Description: The following normal ranges Heart Rate parameters will be used:
  50-90 beats/min
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
beats/min
  screening | 62.2 (8.5) | 67.5 (11.4) | 70.7 (8.6)
  baseline | 63.1 (9.4) | 71 (14) | 71.7 (9.2)
  discharge | 64.9 (7) | 66.9 (10) | 67 (8)

23. Secondary Outcome: Blood Pressure
Description: The following normal ranges Systolic and Diastolic Blood Pressure parameters will be used:
  Systolic Blood Pressure: 100-139 mmHg Diastolic Blood Pressure: 50-89 mmHg
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
mmHg
  Systolic Blood Pressure screening | 120 (12.9) | 126 (21.74) | 121.6 (9.1)
  Systolic Blood Pressure baseline | 116.9 (10.5) | 127.9 (19.7) | 125.5 (14.1)
  Systolic Blood Pressure discharge | 116.9 (10.9) | 124.7 (14.7) | 121.7 (8.9)
  Diastolic Blood Pressure screening | 81.5 (12.1) | 78.9 (11.9) | 80.5 (9.9)
  Diastolic Blood Pressure baseline | 74.5 (10.3) | 79.8 (10.9) | 79.1 (13.3)
  Diastolic Blood Pressure discharge | 75.5 (12.2) | 79 (8.1) | 82 (9.5)

24. Secondary Outcome: SpO2
Description: The following normal ranges SpO2 parameters will be used:
  Peripheral Oxygen Saturation: ≥ 95%
Time Frame: Expected up to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Number analyzed (Participants) | 15 | 15 | 15
percentage
  screening | 99.7 (0.96) | 99.13 (1.25) | 98.53 (1.36)
  baseline | 99.4 (0.91) | 99.13 (0.83) | 98.53 (1.51)
  discharge | 99.33 (0.72) | 99.33 (0.90) | 99 (1.07)

ADVERSE EVENTS:
Time Frame: 7 days
Description: No SAEs and No subject discontinued for AEs
Arm/Group | 3 mL Chloroprocaine HCl 1% | 4 mL Chloroprocaine HCl 1% | 5 mL Chloroprocaine HCl 1%
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 13/15 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mL Chloroprocaine HCl 1% (N=15) | 4 mL Chloroprocaine HCl 1% (N=15) | 5 mL Chloroprocaine HCl 1% (N=15)
Procedural pain (Injury, poisoning and procedural complications) | 14 (17) | 13 (20) | 13 (17) — The most frequent AE was procedural pain (verbatim: pain at the site of surgery)
injection site pain (General disorders) | 2 (2) | 3 (3) | 3 (3)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
diarrhoae (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT02481505/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02481505/SAP_001.pdf